CLINICAL TRIAL: NCT06463145
Title: Effects of a Plant Extract Modulating the Endocannabinoid System and Its Anxiolytic Capacity on Elderly People in Situations of Stress or Anxiety
Brief Title: Study of the Anxiolytic Effects of Aframomum Seed Extract in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nektium Pharma SL (Industry)
Collaborators: Kinetic performance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AME_HCT_2023
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Situational Anxiety
Keywords: Anxiety; Aframomum melegueta seed; Herbal extract; FAAH inhibitor; Quality sleep; Grains of paradise
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the placebo (0 mg) and Botanical extract capsules (50mg, 100mg and 150mg) were identical in appearance to maintain the blindness of the study treatment. Only an unblinded research assistant will have knowledge of which label corresponds to Vanizem doses or placebo. That research assistant will be in charge of: (1) Before each appointment, distributing appropriate treatments or placebo pills into closable pots with a number corresponding to each participant. Care-providers will give closed pots to participants at the time of assessment. (2) Re-labeling all collected data and samples with a participant code number, and sorting into appropriate groups for analysis by blinded researchers.The investigators, study staff, subjects, and statisticians were blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Pill of Food grade Maltodextrin 12 . Once daily for three days.
  Interventions: Dietary Supplement: Placebo
- Vanizem 50mg (Experimental): Pill of Aframomum melegueta extract 50 mg with Food grade Maltodextrin 12 . Once daily for three days.
  Interventions: Dietary Supplement: Vanizem
- Vanizem 100mg (Experimental): Pill of Aframomum melegueta extract 100 mg with Food grade Maltodextrin 12 . Once daily for three days.
  Interventions: Dietary Supplement: Vanizem
- Vanizem 150mg (Experimental): Pill of Aframomum melegueta extract 150 mg with Food grade Maltodextrin 12 . Once daily for three days.
  Interventions: Dietary Supplement: Vanizem

INTERVENTIONS:
Dietary Supplement: Vanizem — Aframomum melegueta seed extract standardized to 10% of total Vanilloid and at least 1.5% of 6-paradol
  Arms: Vanizem 100mg; Vanizem 150mg; Vanizem 50mg
Dietary Supplement: Placebo — Food grade Maltodextrin 12
  Arms: Placebo

SUMMARY:
The goal of this pilot clinical trial is to evaluate if one specific botanical extract from Grains of Paradise works to induce anxiolytic effect in adult people in stress or anxiety situations It will also learn about the extract's positive effects on sleep and mood. The main questions it aims to answer are:

Does botanical extract exert an anxiolytic effect on the participants under stress or anxiety circumstances? Does botanical extract promote positive effects on Mood and nocturnal sleep? Does botanical extract influence body parameters like Blood pressure, inflammatory indicators or stress hormones? Researchers will compare tree doses of botanical extract (50,100 or 150mg) to a placebo (a look-alike substance that contains no herbal product) to see if herbal extract support anxiolytic effect.

Participants will:

Take herbal extract or a placebo daily for 3 days. Visit the clinic two times: at the start of the study (day0) and to the end of the study (Day +2)for checkups and tests.

Keep a diary with questions about their activities, daily foods and physicals perceptions.

DETAILED DESCRIPTION:
The present randomized, double-blind, placebo-controlled crossover trial aims to evaluate the effects of standardized aframomum melegueta seed extract (AME) supplementation on anxiety, mood and sleep quality in healthy men and women experiencing anxious situations. A total of 37 participants were randomly assigned to either AME-first groups or placebo-first group; participants were taken 50, 100 or 150 mg of either AME or matched placebo peels daily for three days. This period is followed by a 1 week washout period at the beginning of which all participants will stop the assigned intervention. After this washout the participants will start their crossover intervention. All Participants were instructed to follow a standardized training program throughout the study, including washout periods to maintain uniformity in physical activity and reduce the effect that exercise can have on stress management. The effects of supplement AME doses compared with a placebo, were evaluated using measures to assess anxiety [The Hamilton Anxiety Scale (HAM-A)], mood [Adapted Profile Mood State (POMS)], sleep quality [Sleep Evaluation Questionnaire (LSEQ) and Pittsburgh Sleep Quality Index (PSQI)]. In addition, some physiological (Blood pressure and heart rate variability), biochemical (minerals, hepatic enzymes and inflammatory biomarkers) and hematological variables (Complete cell count) were determined. Testing was completed at the beginning (Day0) and at the end (Day2) of the supplementation periods with the extract and placebo products to assess acute effects following 3 days of daily use.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 40 and 50 year of age;
* Healthy people with moderate anxiety: HAM-A score in a range between 18 and 24;
* Subject able and willing to participate to the study by complying with the protocol procedures as confirmed by his dated and signed informed consent form;

Exclusion Criteria:

* Score greater than 20 points on the Hamilton Depression Rating Scale (HDRS);
* Receiving medical treatment for anxiety, stress or depression;
* Drugs and alcohol dependence;
* Serious personality disorders that may interfere with participation in the study (psychosis, intense suicidal ideation, etc.);
* In the case of women, having the intention of becoming pregnant;
* Epileptic disorders;
* Liver disorders (cirrhosis, hepatitis, etc.);
* Professional athletes or those who frequently engage in extreme physical activities;
* Impossibility of completing the intervention period due to external factors;

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Anxiety Rating Scale (HAM-A) score | At baseline (day 0) and after intake period (day 2+)
  Change in HAM-A score for Vanizem group compared to placebo control group. 14-items questionnaire reflecting 13 categories of anxiety-related symptom to measure anxiety.

SECONDARY OUTCOMES:
Change in Profile of Mood States (POMS) score | At baseline (day 0) and after intake period (day 2+)
  Change in POMS score for Vanizem group compared to placebo control group. 65-items to evaluate short-term emotional states and represent six subscales assessing tension-anxiety, depression, anger-hostility, fatigue, confusion-bewilderment, and vigor-activity.
Change in Pittsburgh Sleep Quality Index (PSQI) score | At baseline (day 0) and after intake period (day 2+)
  Change in PSQI score for Vanizem group compared to placebo control group. 24-items measuring seven dimensions that can be broadly categorized into sleep efficiency factors (sleep quality, sleep latency, sleep duration, and habitual sleep efficiency) and sleep disturbance factors (sleep disturbance, use of sleep medications, and daytime disturbance).
Change in Leeds Sleep Evaluation Questionnaire (LSEQ) score. 10-items evaluating four domains: ease of initiating sleep, quality of sleep, ease of waking, and behavior following wakefulness. | At baseline (day 0) and after intake period (day 1+ and day 2+)
  Change in LSEQ score for Vanizem group compared to placebo control group.
Change in Heart Rate Variability (HRV) | At baseline (day 0) and after intake period (day 1+ and day 2+)
  Change HRV score for Vanizem group compared to placebo control group. Heart rate variability measured as interbeat intervals (ms) has been collected with POLAR H10+ heart rate bands during sleeping hours.
Change in blood pressure score | At baseline (day 0) and after intake period (day 2+)
  Change in systolic and diastolic blood pressure (mmHg) for Vanizem group compared to placebo control group.
Change in blood cells count | At baseline (day 0) and after intake period (day 2+)
  Changes in a neutrophils, lymphocyte, monocyte, eosinophil, basophil, platelet and red blood cell counts (Cells/mcL) for Vanizem group compared to placebo control group.
Change in blood minerals levels | At baseline (day 0) and after intake period (day 2+)
  Changes in Magnesium (mmol/L) and Zinc (mcmol/L) levels for Vanizem group compared to placebo control group.
Change in blood electrolyte levels | At baseline (day 0) and after intake period (day 2+)
  Changes in Sodium and Chloride levels (mEq/L) for Vanizem group compared to placebo control group.
Change in serum hepatic enzymes | At baseline (day 0) and after intake period (day 2+)
  Changes in gamma-glutamyltransferase (GGT), serum glutamic pyruvic transaminase (GPT), serum glutamic oxaloacetic transaminase (GOT) and alkaline phosphatase (AP) levels (IU/L) for Vanizem group compared to placebo control group.
Change proinflammatory serum biomarkers | At baseline (day 0) and after intake period (day 2+)
  Changes in interleukin-1, interleukin-6, interleukin-8 and tumour necrosis factor alpha levels (pg/mL) for Vanizem group compared to placebo control group.
Change in protein serum biomarker of inflammation | At baseline (day 0) and after intake period (day 2+)
  Changes in c-reactive protein levels (mg/L) for Vanizem group compared to placebo control group.
Change in serum biomarker of stress | At baseline (day 0) and after intake period (day 2+)
  Changes in cortisol (mcg/dL) levels for Vanizem group compared to placebo control group.

OTHER OUTCOMES:
Changes in body composition | At baseline (day 0) and after intake period (day 2+)
  Changes in body fat mass (BFM), body fat percentage (%BF), lean muscle mass (LMM) and percentage of lean muscle mass (%LMM) for Vanizem group compared to placebo control group. Measurements will be assessed using multifrequency bioelectrical impedance analysis (BIA).
Changes in body weight | At baseline (day 0) and after intake period (day 2+)
  Changes in body weight (kg) for Vanizem group compared to placebo control group.
Changes in body mass index (BMI) | At baseline (day 0) and after intake period (day 2+)
  BMI for Vanizem group compared to placebo control group. Weight (kg) and height (cm) will be combined to report BMI in (kg/cm^2).

CONTACTS AND LOCATIONS:
Overall Officials: Laura López-Rios, PhD, Principal Investigator — Nektium Pharma SL
Locations (1):
- Kinetic perfomance SL, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Umukoro S. and Aladeokin A. C., Therapeutic effects of grains of paradise (aframomum melegueta) seeds Nuts and Seeds in Health and Disease Prevention, 2011, Academic Press, Cambridge, MA, USA, 535-543.
- [Background] Ilic NM, Dey M, Poulev AA, Logendra S, Kuhn PE, Raskin I. Anti-inflammatory activity of grains of paradise (Aframomum melegueta Schum) extract. J Agric Food Chem. 2014 Oct 29;62(43):10452-7. doi: 10.1021/jf5026086. Epub 2014 Oct 20. PMID 25293633
- [Background] Ogwu, M.C., Dunkwu-Okafor, A., Omakor, I.A., Izah, S.C. (2024). Medicinal Spice, Aframomum melegueta: An Overview of the Phytochemical Constituents, Nutritional Characteristics, and Ethnomedicinal Values for Sustainability. In: Izah, S.C., Ogwu, M.C., Akram, M. (eds) Herbal Medicine Phytochemistry. Reference Series in Phytochemistry. Springer, Cham. https://doi.org/10.1007/978-3-031-21973-3_72-1
- [Background] Umukoro S, Ashorobi RB. Further studies on the antinociceptive action of aqueous seed extract of Aframomum melegueta. J Ethnopharmacol. 2007 Feb 12;109(3):501-4. doi: 10.1016/j.jep.2006.08.025. Epub 2006 Sep 3. PMID 17023130
- [Background] Ford JL, Ildefonso K, Jones ML, Arvinen-Barrow M. Sport-related anxiety: current insights. Open Access J Sports Med. 2017 Oct 27;8:205-212. doi: 10.2147/OAJSM.S125845. eCollection 2017. PMID 29138604
- [Background] Halson SL, Juliff LE. Sleep, sport, and the brain. Prog Brain Res. 2017;234:13-31. doi: 10.1016/bs.pbr.2017.06.006. Epub 2017 Jul 17. PMID 29031461
- [Background] Patel S, Hill MN, Cheer JF, Wotjak CT, Holmes A. The endocannabinoid system as a target for novel anxiolytic drugs. Neurosci Biobehav Rev. 2017 May;76(Pt A):56-66. doi: 10.1016/j.neubiorev.2016.12.033. PMID 28434588
- [Background] Batista LA, Gobira PH, Viana TG, Aguiar DC, Moreira FA. Inhibition of endocannabinoid neuronal uptake and hydrolysis as strategies for developing anxiolytic drugs. Behav Pharmacol. 2014 Sep;25(5-6):425-33. doi: 10.1097/FBP.0000000000000073. PMID 25083569